CLINICAL TRIAL: NCT04371445
Title: Intracanalicular Dexamethasone Insert for Management of Post-operative Pain and Inflammation in Patients Undergoing Vitreoretinal Surgery
Brief Title: Dextenza in the Post-op Management of Vitreoretinal Surgeries
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Principal Investigator, Katherine Talcott, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4-29-2020
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Vitreoretinal Surgery; Ocular Inflammation; Post-operative Pain; Post-Operative Inflammation
Keywords: dexamethasone insert; Ocular Inflammation; Post-Operative Inflammation; Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Calcium Dobesilate; prednisolone acetate; Methylprednisolone

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Only the readers of the anterior segment OCT will be masked.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intracanalicular dexamethasone insert group (Experimental): This arm will receive the DEXTENZA® insert within minutes after the completion of the surgery.
  Interventions: Drug: Dexamethasone Ophthalmic Insert
- Topical steroid drop group (Active Comparator): This arm will receive the prescription for daily prednisolone acetate 1% eye drops 4 times a day for the first week following the procedure, starting on the day of surgery.
  Interventions: Drug: Prednisolone Acetate 1% Oph Susp

INTERVENTIONS:
Drug: Dexamethasone Ophthalmic Insert — DEXTENZA® is a 3mm long gel-like cylinder that is inserted in the punctum, a natural opening in the lower eyelid. DEXTENZA® is activated by the eye's moisture. DEXTENZA® delivers 0.4 mg dexamethasone, a liquid corticosteroid, onto the surface of the eye automatically for up to 30 days after eye surgery. Dexamethasone is used to reduce inflammation and eye pain. This arm will also receive the standard of care topical ofloxacin eye drop antibiotic regimen.DEXTENZA® is a 3mm long gel-like cylinder that is inserted in the punctum, a natural opening in the lower eyelid. DEXTENZA® is activated by the eye's moisture. DEXTENZA® delivers 0.4 mg dexamethasone, a liquid corticosteroid, onto the surface of the eye automatically for up to 30 days after eye surgery. Dexamethasone is used to reduce inflammation and eye pain. This arm will also receive the standard of care including topical antibiotics.
  Other Names: DEXTENZA®
  Arms: Intracanalicular dexamethasone insert group
Drug: Prednisolone Acetate 1% Oph Susp — Prednisolone acetate 1% eye drops are used 2-4 times daily for 30 days as the current standard of care for treating inflammation and eye pain after cataract surgery. Prednisolone, like dexamethasone, is a steroid. This arm will also receive the standard of care including topical antibiotics.
  Other Names: PRED FORTE®, OMNIPRED®
  Arms: Topical steroid drop group

SUMMARY:
This study will assess the control of inflammation at days 1, 7, 14, and 21 days following the vitreoretinal surgical procedure analyzing two randomized study arms: Intracanalicular dexamethasone insert group or topical steroid drop group.

Patients must be 18 years of age and older, of any race and either sex, requiring surgery with the procedure type of pars plana vitrectomy for either the indication of macular hole, epiretinal membrane removal, or vitreomacular traction.

DETAILED DESCRIPTION:
Topical steroids are the current standard of care for managing postoperative pain and inflammation following vitreoretinal surgery. However, topical treatments are limited by the potential for patient non-adherence and variation in drug concentrations due to the intermittent nature of application. A corticosteroid insert, placed following surgery, provides the advantages of reliable and continuous drug delivery without the need for patients to adhere to a treatment regimen. Recently, DEXTENZA®, a dexamethasone intracanalicular insert was FDA-approved for the treatment of inflammation and pain following ophthalmic surgery. DEXTENZA® is placed into the canaliculus via the lower punctum and is designed to release steroid medication for 30 days.

The data is limited regarding the safety and efficacy of DEXTENZA® for postoperative management of vitreoretinal surgery. Herein, the aim of this study is to assess the management of pain and inflammation following retinal surgery when using a dexamethasone implant compared with topical steroids.

ELIGIBILITY:
Inclusion Criteria:

* Men and women >18 years old
* Planning to undergo vitreoretinal surgery with the procedure type of pars plana vitrectomy for either the indication of macular hole, epiretinal membrane removal, or vitreomacular traction.

Exclusion Criteria:

* Patients undergoing combined cataract or glaucoma procedure, intraocular lens exchange, scleral buckle, and/or implant of a drug delivery system
* History of complications, trauma, adverse events, disease in nasolacrimal region, including dacryocystitis, canaliculitis in either eye
* Structural lid abnormalities such as ectropion or entropion in surgical eye
* Ongoing use of systemic narcotic pain relievers
* Presence of any intraocular inflammation (cells and flare) in the study eye at screening/baseline
* Pain score greater than "0" on the ocular pain assessment in the study eye at screening/baseline
* Active or chronic or recurrent uncontrolled ocular or systemic inflammatory disease, including diabetes
* Other ocular surgeries or procedures during the study period and/or 6 months prior
* Intraoperative complications
* Patients with history of glaucoma (defined as glaucoma requiring 2 or more drops, IOP at baseline greater than 25, or advanced optic nerve cupping). Patients with glaucoma or ocular hypertension controlled with a single drop can be enrolled.
* Patients with a known hypersensitivity to NSAIDs or steroids or any component of the study medication.
* Have used ocular, topical, or systemic NSAIDs within 7 days prior to procedure and during surgery.
* Use of intracameral or subconjunctival NSAIDs or steroids intraoperatively.
* Have used topical, ocular, inhaled or systemic steroids within 14 days prior to procedure
* Are pregnant or nursing/lactating
* Participation as a subject in any clinical study within the 30 days prior to randomization.
* Surgeries using 20 gauge or 23 gauge instruments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
To assess control of inflammation following the vitreoretinal surgical procedure. | day 14 following surgery
  Percentage of patients with Inflammation following surgery as assessed from 0-4+ cell and flare based on the Standardization of Uveitis Nomenclature [SUN] Working Group grading scheme at day 14

SECONDARY OUTCOMES:
The patient reporting of pain following surgery using visual analog pain scale at days 1, 3, 7, 14, and 21 following surgery. | days 1, 3, 7, 14, and 21 following surgery
  Pain following surgery will be measured using a scale from 0 to10 (0 = no pain, 10 = severe pain that prevents performing activities of daily living). Higher scores mean a worse outcome.
Inflammation assessed on Anterior Segment OCT by masked grading at days 1, 7, 14, and 21 following surgery. | days 1, 7, 14, and 21 following surgery
  Anterior segment will be assessed using a continuous variable (cells/mm3).
Mean change in Best Corrected Visual Acuity (BCVA) from baseline to day 21 following surgery. | day 21 following surgery
  BCVA was assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) method.
% of patients with rebound inflammation defined as a two-step worsening of inflammation by SUN grading. | day 21 following surgery
% of patients receiving rescue treatment. | days 1, 7, 14, and 21 following surgery
% of patients with postoperative management via telephone or electronic messaging | day 21 following surgery
The incidence and severity of ocular and non-ocular adverse events (AEs) and serious AEs between arms. | day 21 following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Talcott, M.D., Principal Investigator — Cole Eye Institute, Cleveland Clinic
Locations (1):
- Cole Eye Institute, Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Hermann MM, Ustundag C, Diestelhorst M. Electronic compliance monitoring of topical treatment after ophthalmic surgery. Int Ophthalmol. 2010 Aug;30(4):385-90. doi: 10.1007/s10792-010-9362-3. Epub 2010 Apr 7. PMID 20373127
- [Background] An JA, Kasner O, Samek DA, Levesque V. Evaluation of eyedrop administration by inexperienced patients after cataract surgery. J Cataract Refract Surg. 2014 Nov;40(11):1857-61. doi: 10.1016/j.jcrs.2014.02.037. Epub 2014 Sep 22. PMID 25248295
- [Background] Tyson SL, Bafna S, Gira JP, Goldberg DF, Jones JJ, Jones MP, Kim JK, Martel JM, Nordlund ML, Piovanetti-Perez IK, Singh IP, Metzinger JL, Mulani D, Sane S, Talamo JH, Goldstein MH; Dextenza Study Group. Multicenter randomized phase 3 study of a sustained-release intracanalicular dexamethasone insert for treatment of ocular inflammation and pain after cataract surgery. J Cataract Refract Surg. 2019 Feb;45(2):204-212. doi: 10.1016/j.jcrs.2018.09.023. Epub 2018 Oct 24. PMID 30367938
- [Background] Gira JP, Sampson R, Silverstein SM, Walters TR, Metzinger JL, Talamo JH. Evaluating the patient experience after implantation of a 0.4 mg sustained release dexamethasone intracanalicular insert (Dextenza): results of a qualitative survey. Patient Prefer Adherence. 2017 Mar 8;11:487-494. doi: 10.2147/PPA.S126283. eCollection 2017. PMID 28331295
- [Background] Jabs DA, Nussenblatt RB, Rosenbaum JT; Standardization of Uveitis Nomenclature (SUN) Working Group. Standardization of uveitis nomenclature for reporting clinical data. Results of the First International Workshop. Am J Ophthalmol. 2005 Sep;140(3):509-16. doi: 10.1016/j.ajo.2005.03.057. PMID 16196117